CLINICAL TRIAL: NCT06176222
Title: To Investigate the Effects of Combined Use of Naldebain® ER Injection and Precedex® After Video-assisted Thoracoscopic Surgery
Brief Title: Combined Use of Naldebain® ER Injection and Precedex® After VATS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20230150
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-10

CONDITIONS: Acute Post Operative Pain; Chronic Post Operative Pain; Postoperative Complications
Keywords: Multimodal Analgesia; Dinalbuphine Sebacate; Dexmedetomidine; Video-Assisted Thoracic Surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Precedex Group (Experimental): Drug: PRECEDEX INJ★ 2ML Dosage form: 100 mcg/ml dexmedetomidine Dosage: 0.1~0.4 mcg/kg/hr intravenous infusion Frequency and Duration: intrvenous infusion 12 hours after the surgery immediately
  Interventions: Drug: PRECEDEX INJ★ 2ML
- Placebo Group (Placebo Comparator): Drug: 0.9% Normal Sline Dosage: 0.1 ml/kg/hr intravenous infusion Frequency and Duration: intrvenous infusion 12 hours after the surgery immediately
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: PRECEDEX INJ★ 2ML — patient received PRECEDEX INJ★ 2ML 0.1~0.4 mcg/kg/hr intravenous infusion 12 hours after the surgery immediately
  Other Names: Dexmedetomidine
  Arms: Precedex Group
Drug: Normal saline — patient received Normal Saline 0.1 ml/kg/hr intravenous infusion 12 hours after the surgery immediately
  Other Names: 0.9% Normal Saline
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to investigate the effects of combined use of Naldebain® ER Injection and Precedex® in patients received video-assisted thoracoscopic surgery. The main questions it aims to answer are:

* the pain intensity after surgery
* the level of dizziness after surgery Participants will receice ultrasound-guided thoracic paravertebral nerve block, intramuscular Naldebain® ER injection and intravenous Precedex® infusion.

If there is a comparison group: Researchers will compare experimental group with placebo group to see if pain and dizziness after surgery can reduced.

DETAILED DESCRIPTION:
Ⅰ.Protocol title: To investigate the effects of combined use of Naldebain® ER Injection and Precedex® after video-assisted thoracoscopic surgery

Ⅱ.Objectives: Video-assisted thoracoscopic surgery (VATS) is currently the mainstream of thoracic surgery, but it may also cause stronger postoperative pain than expected. Therefore, pain control after thoracoscopic surgery is very important, because increased acute pain will increase the incidence of chronic pain, and untreated pain may lead to increased postoperative complications. At present, the combined use of regional nerve block, opioids, and non-steroidal anti-inflammatory drugs is the current mainstream strategy for multimodal analgesia after thoracoscopic surgery.

Paravertebral block (PVB) involves injecting a local anesthetic into the paravertebral wedge-shaped space as it emerges from the intervertebral foramen. It produces an ipsilateral somatosensory and sympathetic block, and has good analgesic effects on anesthesia and unilaterally induced pain from the chest and abdomen. So far, thoracic paravertebral block (TPVB) is considered the best alternative to thoracic epidural analgesia because it can provide effective immediate postoperative analgesic effect in patients undergoing VATS.

Naldebain® ER Injection is a long-acting prodrug of Nalbuphine, aimed at addressing the medical need for long-acting analgesics. It is an agonist-antagonist of synthetic phenanthrene series opioids. It is chemically related to the widely used opioid antagonist naloxone and the potent opioid pain reliever oxymorphone. At present, nalbuphine sebacate has been used in many surgical procedures to relieve postoperative pain.

Precedex® injection (dexmedetomidine hydrochloride), a centrally acting α2-receptor agonist, has the same sedative effects as other benzodiazepine drugs. However, due to the different pharmacological mechanisms, there are no side effects such as respiratory depression and delirium. In addition, according to Venn et al. in 2000, when 33 postoperative patients were using respirators in the intensive care unit, they found that the use of dexmedetomidine could reduce the use of morphine by 50%, thereby reducing the possible side effects of opioids and as a good adjuvant drug for pain relief.

In view of the fact that patients undergo thoracoscopic surgery, good analgesic function is crucial for the recovery of postoperative pulmonary function. Therefore, the purpose of this study is to investigate the application effect of the multimodal analgesic formula combined with thoracic paravertebral nerve block, Naldebain® ER Injection and Precedex® injection after VATS.

III. Study design 1. ☑ Control: ☑ placebo

* active (please specify name and dosage)

  * others
  * Uncontrolled 2. Blinding: □ open-label □ single blind ☑ double blind □ others 3. Randomized: ☑ yes □ no 4. ☑ Parallel □ cross-over □ others 5. Duration of study：from IRB approval ~to 2025 , 12 , 31 ,total 24 months Duration of Enrollment : from IRB approval ~to 2025 , 12 , 31 ,total 24 months Duration of treatment：from IRB approval ~to 2025 , 12, 31 ,total 24 months Duration of follow-up: from IRB approval ~to 2025 , 12 , 31 ,total 24 months
  * Multi-national □multi-center(Taiwan) ☑single center(Taiwan) 6. Number of subjects: 70 7. Is there any of the followings included DSMB, Data Safety Monitoring Board:
  * yes ☑ no IV. Assessment criteria

    1. Efficacy:

       It can effectively reduce the expected moderate and severe acute pain after surgery, and reduce the degree and incidence of side effects of analgesic drugs.
    2. Safety:

       Side Effects: Hypotension, hypertension, nausea, bradycardia, fever, vomiting, tissue hypoxia, tachycardia, and anemia.

       Contraindications: Dexmedetomidine Hydrochloride is contraindicated in patients who are known to be allergic to the components of Dexmedetomidine.

       Precautions: 1. For patients with severe heart block and/or severe ventricular insufficiency, it should be used with caution. Since Precedex reduces the activity of sympathetic nerves, it can be expected that the effect of hypotension and/or bradycardia may be more pronounced in patients with low blood volume, diabetes or chronic hypertension, and elderly patients. 2. When it is necessary to use other vasodilators or drugs that lower the heart rate (negative chronotropic agents), administering Precedex at the same time may have a drug effect and should be used with caution.

       Overdose: Discontinue immediately. Oxygen, intravenous drips, vasoconstrictors, and other supportive therapies may be used as needed.

       V. Selection criteria

    <!-- -->

    1. Main inclusion criteria:

    <!-- -->

    1. Subject's age: 20~65 years old
    2. ASA classification: I~III
    3. Patients who need postoperative pain relief due to thoracoscopic surgery 2. Main exclusion criteria: 1. The patient suffers from a communication disorder 2. The patient has coagulopathy 3. Sick with obvious heart, lung, liver or kidney disease 4. The patient's body mass index is less than 18.5 or greater than 35 5. Pregnant patients 6. Patients who took opioids for more than three weeks before surgery 7. Patients with contraindications to local anesthesia 8. Patients with a history of chronic pain 9. Patients with a history of drug allergy to Naldebain® ER Injection, COX2-inhibitor NSAIDs (such as parecoxib), or Precedex® VI. Statistical analysis

    <!-- -->

    1. Statistical Method for Efficacy / Safety measurements:

The basic characteristics of the two groups of patients are presented with descriptive statistics. All results are expressed as mean ± standard deviation (SD) or applicable percentage. The differences between the groups were analyzed using ANOVA (one-way analysis of variance), and then paired comparisons were made with the post-event Student-Newman-Keuls-Test. The classified data is analyzed using X2 or Fisher's exact test. P value less than 0.05 is considered to be a significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age: 18~65 years old
2. ASA classification: I~III Exclusion Criteria:
3. Patients who need postoperative pain relief due to thoracoscopic surgery

Exclusion Criteria:

1. The patient suffers from a communication disorder
2. The patient has coagulopathy
3. Sick with obvious heart, lung, liver or kidney disease
4. The patient's body mass index is less than 18.5 or greater than 35
5. Pregnant patients
6. Patients who took opioids for more than three weeks before surgery
7. Patients with contraindications to local anesthesia
8. Patients with a history of chronic pain
9. Patients with a history of drug allergy to Naldebain® ER Injection, COX2-inhibitor NSAIDs (such as parecoxib), or Precedex®

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-28 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
poatoperative analgesic effect | During the 60 minutes of rest in the PACU, the patient's pain intensity was assessed every fifteen minutes.
  Use the numerical rating scale (NRS) score to ass the intensity of pain after surgery
poatoperative analgesic effect | the first morning and afternoon after surgery, and the second morning and afternoon after surgery
  Use the numerical rating scale (NRS) score to ass the intensity of pain after surgery
poatoperative analgesic effect | the third day after surgery, the fourth day after surgery, the fifth day after surgery, and the sixth day after surgery
  Use the numerical rating scale (NRS) score to ass the intensity of pain after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, MD, PhD, Principal Investigator — Department of anesthesiology, Kaohsiung Medical University Hospital
Locations (1):
- Hung-Te Hsu, Kaohsiung City, Taiwan